CLINICAL TRIAL: NCT02436811
Title: Literacy and Information Retention in Pregnancy
Brief Title: Oral Health Literacy and Oral Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Paraná (Other)
Responsible Party: Principal Investigator, Luciana Reichert Assunção Zanon, Adjunct Professor, Universidade Federal do Paraná
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CAAE 27273314.1.0000.0102
Record Dates: First submitted 2015-04-29; First posted 2015-05-07 (Estimated); Results first posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-04

CONDITIONS: Retention
Keywords: Health literacy; Pregnant women; Feeding behaviour; Oral health; Child
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standardized oral instruction (Experimental): 60 women aged between 12 and 50 and gestational period of up to 32nd weeks. A trained individual will present the same information arranged in the educational brochure in the intervention group on standardized oral form. This examiner will be trained in a unified way in relation to the instructions available in the form of written guidance. Thus, the only difference between the two measures is the interaction between the participant and researcher orally.
  Interventions: Behavioral: Written form instruction; Behavioral: Control
- Written form instruction (Experimental): 60 women aged between 12 and 50 and gestational period of up to 32nd weeks. Participants in writing intervention will receive a brochure containing information on diet and oral health. This leaflet was produced in accordance with the recommendations of the Ministry of Health regarding eating habits for children under two years (BRAZIL, 2002) and according to the Health Book of the Child: Growth and Development (BRAZIL, 2012).
  Interventions: Behavioral: Standardized oral instruction; Behavioral: Control
- Control (Experimental): 60 women aged between 12 and 50 and gestational period until 32nd weeks.The control group will receive a leaflet on oral cancer.
  Interventions: Behavioral: Written form instruction; Behavioral: Standardized oral instruction

INTERVENTIONS:
Behavioral: Written form instruction — 60 women aged between 12 and 50 and gestational period of up to 32nd weeks. Participants in writing intervention will receive a brochure containing information on diet and oral health. This leaflet was produced in accordance with the recommendations of the Ministry of Health regarding eating habits for children under two years (BRAZIL, 2002) and according to the Health Book of the Child: Growth and Development (BRAZIL, 2012).
  Arms: Control; Standardized oral instruction
Behavioral: Standardized oral instruction — 60 women aged between 12 and 50 and gestational period of up to 32nd weeks. A trained individual will present the same information arranged in the educational brochure in the intervention group on standardized oral form. This examiner will be trained in a unified way in relation to the instructions available in the form of written guidance. Thus, the only difference between the two measures is the interaction between the participant and researcher orally.
  Arms: Control; Written form instruction
Behavioral: Control — 60 women aged between 12 and 50 and gestational period until 32nd weeks.The control group will receive a leaflet on oral cancer.
  Arms: Standardized oral instruction; Written form instruction

SUMMARY:
This is study aims to evaluate the retention of information on oral health and eating habits in children under two years of age. A total of 180 pregnant women aged between twelve and fifty years of age will be selected for this study. Before the randomization process, the literacy in oral health score will be assessed through previously validated instrument BREALD- 30. Participants will be randomly selected according to the value of BREALD-30, categorized as adequate (≥18) and low (<18) in a specific intervention. Interventions occur in written form through an educational brochure or standardized oral, both with information about the feeding practices and oral health in children under two years. The control group will be the implementation of an educational booklet on oral cancer. To evaluate the association between variables pregnant women will respond to a semi-structured form with questions regarding oral health and nutrition, in three different times: before the intervention, 15 minutes after the intervention and 4 weeks after the intervention. Social and economic and demographic data will be evaluated at baseline. The data will be statistically analyzed by Student's t-tests and ANOVA paired, adopting a 5% significance level. In the event of non-normality of the data, the corresponding non-parametric statistical tests will be applied. This study has the hypothesis that the written intervention presents best results in participants with high literacy and the standardized oral with those with low literacy.

DETAILED DESCRIPTION:
This study has the objective to verify the relationship between oral health literacy and information retention in health in pregnant women.

A total of 180 pregnant women with age between 12 and 50 years will be recruited to participate in this study. The inclusion criteria are: gestational age up to 32 weeks and who do not have any health problems that would prohibit participation in the study.

In a first moment, the instrument BREALD-30 (Brazilian Rapid Estimate of Adult Literacy in Dentistry), validated for Brazilian portuguese, will be applied to pregnant women who accept to participate voluntarily in the study . This instrument is composed of 30 words related to oral health. These words should be read aloud to the interviewer, each word read correctly, will receive a score equivalent to 1 (one). Thus, the scores can range from 0 (lowest literacy) to 30 (highest literacy). Pregnant women will be classified according to the score achieved in appropriate literacy (equal and more than 18 points) and low literacy (lower than 18 points) according to the value obtained in the lowest quintile. The reading of the instrument's words lasts about two minutes.

After applying the BREALD-30 instrument, the pregnant women will receive a previously tested form with social and economic and demographic information. This information includes maternal age, marital status (categorized into single, married, separated and widow), number of children, occupation and family income. It will be included a list of household items for assessment of social and economic results according to the criteria of the Brazilian Association of Research Companies.

It will be also assessed the degree of knowledge of mothers about feeding habits and oral health of children under two years of age. This step will include the establishment of a list of statements that express opinions with variations in responses: agree, neither agree nor disagree, disagree and do not know, in a Likert scale. The answers are scored 0-1. Scores can vary from 0 to 9. The application form will last about 10 minutes.

According to the results of BREALD-30, pregnant women will be randomly selected to receive an educational intervention, which is related to oral health and feeding habits in children under two-years of age. After enrollment, the participants will be randomized (1: 1: 1) in three groups: written instruction, oral instruction and control, by raffle using sealed, opaque envelopes. Each group will consist of 60 participants.

Group writing intervention: 60 women aged between 12 and 50 and gestational period of up to 32nd weeks. Participants in writing intervention will receive a brochure containing information on diet and oral health. This leaflet was produced in accordance with the recommendations of the Ministry of Health regarding eating habits for children under two years (BRAZIL, 2002) and according to the Health Book of the Child: Growth and Development (BRAZIL, 2012).

Group oral intervention: 60 women aged between 12 and 50 and gestational period of up to 32nd weeks. A trained individual will present the same information arranged in the educational brochure in the intervention group on standardized oral form. This examiner will be trained in a unified way in relation to the instructions available in the form of written guidance. Thus, the only difference between the two measures is the interaction between the participant and researcher orally.

Control group: 60 women aged between 12 and 50 and gestational period until 32nd weeks.The control group will receive a leaflet on oral cancer.

After the educational guidelines pregnant women will respond the same form applied before the interventions, with questions about the relationship between oral health and eating habits in children under two years of age.

Four weeks after the first procedure the same form will be reapplied to assess the retention of health knowledge after an interval of time.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* To be literate
* Pregnancy maximum in the 32nd week

Exclusion Criteria:

* Physical or mental disability

Ages: 12 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 180 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luciana R Zanon, DDS, Principal Investigator — Adjunct professor
Locations (1):
- Karina Duarte Vilella, Curitiba, Brazil, Brazil

RESULTS

PARTICIPANT FLOW:
Groups:
- Standardized Oral Instruction: women aged between 12 and 50 and gestational period of up to 32nd weeks. A trained individual will present the same information arranged in the educational brochure in the intervention group on standardized oral form. This examiner will be trained in a unified way in relation to the instructions available in the form of written guidance. Thus, the only difference between the two measures is the interaction between the participant and researcher orally.
- Written Form Instruction: women aged between 12 and 50 and gestational period of up to 32nd weeks. Participants in writing intervention will receive a brochure containing information on diet and oral health. This leaflet was produced in accordance with the recommendations of the Ministry of Health regarding eating habits for children under two years (BRAZIL, 2002) and according to the Health Book of the Child: Growth and Development (BRAZIL, 2012).
- Control: women aged between 12 and 50 and gestational period until 32nd weeks.The control group will receive a leaflet on oral cancer.
Period: Overall Study
Arm/Group | Standardized Oral Instruction | Written Form Instruction | Control
Started | 60 | 60 | 60
Completed | 58 | 51 | 53
Not Completed | 2 | 9 | 7
Not completed — Lost to Follow-up | 2 | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standardized Oral Instruction | Written Form Instruction | Control | Total
Number analyzed (Participants) | 60 | 60 | 60 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 12 | 8 | 32
  Between 18 and 65 years | 48 | 48 | 52 | 148
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.60 (5.74) | 26.32 (6.19) | 25.58 (6.59) | 26.22 (6.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 60 | 60 | 180
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 60 | 60 | 60 | 180

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Knowledge Score
Description: The knowledge score was assessed by nine statements developed and tested in a pilot study including items related to breastfeeding, supplemental feeding, sugar intake, bottle use, oral hygiene, and use of fluoride toothpaste. These statements were rated on a three-level Likert scale, under the following options: "agree," "neither agree nor disagree," and "disagree," in addition to "I don't know." Each correct answer received score 1 whereas incorrect answers such as "neither agree nor disagree" and "I don't know" were assigned score 0. The final scores ranged from 0 to 9. Higher values indicate better outcomes.
Time Frame: The nine statements were applied before the intervention (pre-test), after a 15-minute break, the statements were applied again (post-test). After a 4-week interval, the statement were applied once again.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standardized Oral Instruction | Written Form Instruction | Control
Number analyzed (Participants) | 58 | 51 | 53
units on a scale
  Pre-test | 4.81 (1.45) | 4.86 (1.56) | 4.64 (1.39)
  Post-test | 7.10 (1.52) | 5.84 (1.73) | 4.74 (1.58)
  4-week interval | 6.34 (1.45) | 5.41 (1.56) | 4.83 (1.38)
Statistical Analysis 1: Comparison: Standardized Oral Instruction vs Written Form Instruction vs Control; Univariate and multivariate Poisson regressions with robust variance were obtained to estimate the rate ratios (RR) and their respective 95% confidence intervals. Two Poisson regression models were generated, using the knowledge score 15 minutes after the intervention (post-test) and 4 weeks after the interventions (follow-up test) as dependent variables; Test type: Superiority or Other; p < 0.001, Regression, Poisson — A stepwise forward selection model was used. All independent variables with P<0.20 in the univariate analysis were selected and those which were significant (P<0.05) were kept in the final model. The level of significance was 5%

ADVERSE EVENTS:
Time Frame: 1 month
Description: The total number of "0" of participants at risk means that no serious adverse events were assessed as this study aimed to verify the gain of information in oral health during the follow-up period.
Arm/Group | Standardized Oral Instruction | Written Form Instruction | Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standardized Oral Instruction (N=0) | Written Form Instruction (N=0) | Control (N=0)
knowledge score variation (Social circumstances) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standardized Oral Instruction (N=0) | Written Form Instruction (N=0) | Control (N=0)
knowledge score variation (Social circumstances) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes